CLINICAL TRIAL: NCT04845984
Title: Evaluation of the Prevalence of SARS-CoV-2 Infection in the Healthcare Workers (HCWs) in Five Hospital of the Alpine Region
Brief Title: Evaluation of the Prevalence of SARS-CoV-2 Infection in the Healthcare Workers (HCWs) in Four Hospital of the Alpine Region
Acronym: PACAAP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Other Study IDs: 20-12
Record Dates: First submitted 2021-03-02; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Health Care Worker
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PACAAP study aims to report the seroprevalence of SARS-CoV-2 IgG antibodies among HCWs testing during the massive campaign screening set up in France by French ministry of Health and national authorities in four hospital of the Alpine region.

DETAILED DESCRIPTION:
In France during the first wave of the pandemic, 30,230 symptomatic healthcare workers had been reported positive. Yet, the prevalence of the infection in French healthcare workers remains unknown as it mostly reflect symptomatic infections.

Also, the prevalence of infection was reported being higher in male healthcare workers, and in those having patients' facing roles. However, the impact of the level of exposure to SARS-CoV-2, the use of personal protective equipment and hospital organization to prevent infection and spread remains unclear.

Our study aims to report the seroprevalence of SARS-CoV-2 infection among French healthcare workers after the first wave of the pandemic. It also aims to explore the impact of the type of occupations and the level of exposure to the viruses on the seroprevalence of infection.

ELIGIBILITY:
Inclusion Criteria:

* Hospital staff employee
* Employed in one of the participating centers
* Volunteers to perform SARS-CoV-2 serology
* Permanent or occasional staff (temporary workers, short contracts)
* Caregivers or not (medical, paramedical, administrative, technical staff)

Exclusion Criteria:

* Staff who are not working at a participating center while participating in the study
* Person under guardianship or curatorship
* Opposition to data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be proposed to all the staff of participating hospitals, who have been tested for SARS-CoV-2 (serology) and who have not objected to the use of their health data.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 prevalency among hospital health care professionals | Day 1
  Number of Health Care Worker with an antibody test (IgG) positive for SARS-CoV2

CONTACTS AND LOCATIONS:
Locations (1):
- Ch Annecy Genevois, Pringy, France

IPD SHARING:
Plan to Share IPD: No